CLINICAL TRIAL: NCT06299423
Title: Perioperative Electrocardiogram Remote Monitoring to Assess Preoperative Psychological Distress and Improve Postoperative Recovery in Inflammatory Bowel Disease Surgery: a Pilot Single-arm Prospective Study
Brief Title: Perioperative Monitoring to Assess Preoperative Anxiety in Inflammatory Bowel Disease Patients
Acronym: PeRseo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 3677
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Inflammatory Bowel Diseases; Surgery
Keywords: Inflammatory Bowel Disease; Surgery; Anxiety and Depression
MeSH Terms: conditions — Inflammatory Bowel Diseases; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Single-center, interventional, case-series study with a historical cohort of comparison
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Howdy Senior® device (Experimental): Patients will undergo standard perioperative management. Additionally, patients will perform three preoperative and twelve postoperative HOWDY Senior® assessments. The assessment consists of a nocturnal electrocardiogram (ECG) measure and a morning rest Heart Rate Variability (HRV) measure of five minutes.
  Interventions: Device: Howdy Senior® device
- Standard perioperative management (No Intervention): Patients belonging to the historical cohort of comparison, who underwent standard perioperative management and surgical intervention between January 2021 and January 2022.

INTERVENTIONS:
Device: Howdy Senior® device — Standard perioperative management plus three preoperative and twelve postoperative (until 90 days after surgery) HOWDY Senior® device assessments.
  Arms: Howdy Senior® device

SUMMARY:
Anxiety and depression are extremely common among Inflammatory Bowel Disease (IBD) patients undergoing surgery and may increase the risk of postoperative adverse outcomes. This study aims to objectively evaluate preoperative psychological distress by remotely measuring the patient's physiological parameters and Heart Rate Variability (HRV) with the Howdy Senior ® device (Comftech Srl). Additionally, the study will also investigate the feasibility and effectiveness of the Howdy Senior® device in improving the postoperative patient's monitoring.

DETAILED DESCRIPTION:
Inflammatory Bowel Disease (IBD) patients are at high risk of postoperative complications and delayed recovery. Preoperative anxiety and low patient's awareness of the disease may increase the risk of postoperative complications inducing an autonomic impairment which may in turn determine an inflammatory unbalance. This correlation can be confirmed through the preoperative monitoring of the autonomic function- with wearable electrocardiogram (ECG) devices. The Howdy Senior® device (ComfTech Srl) allows the real-time remote ECG monitoring and the computation of stress and fatigue indexes.

The Howdy Senior® device may also provide a reliable tool for remotely monitoring the patient's clinical parameters after discharge.

This study aims to explore the pathophysiological mechanisms linking preoperative anxiety and autonomic response and assess the feasibility and effectiveness of the Howdy Senior® device for the postoperative patients' remote monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged more than 18 years old.
* Established Crohn's disease (CD) or Ulcerative Colitis (UC) at the time of surgery indication with a proven histological diagnosis.
* Patients scheduled for elective intestinal resection.

Exclusion Criteria:

* Diagnosis of Undetermined Colitis.
* Recurrent disease.
* Concomitant diagnosis of malignancy.
* Established diagnosis of major depressive disorder or anxiety disorder.
* Diagnosis of ventricular or supraventricular arrythmia.
* Active pharmacological treatment with β-blockers or other drugs affecting the heart rate.
* Known hypersensitivity to cotton or silver.
* Emergent surgery.
* Planned open surgery.
* Any concomitant surgery unrelated to the main surgical indication. Patients undergoing perianal surgery for related perianal disease can be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between preoperative anxiety and preoperative Heart Rate Variability (HRV) | From 14 days to 1 day before surgery
  Correlation between preoperative anxiety- assessed through the Hospital Anxiety and Depression Scale (HADS) (Self-reporting scale ranging from 0 to 21, where significant anxiety and depression are identified by a 8 point cut-off) and the median value of at least three Heart Rate Variability (HRV) measures collected in the preoperative period through the Howdy Senior® device.

SECONDARY OUTCOMES:
Correlation between preoperative anxiety and 90-day Comprehensive Complication Index (CCI) | 90 days after surgery
  Correlation between preoperative anxiety- assessed through the Hospital Anxiety and Depression Scale (HADS) (Self-reporting scale ranging from 0 to 21, where significant anxiety and depression are identified by a 8 point cut-off) and the median value of the Comprehensive Complication Index (CCI) (Index ranging from 0 (no complication) to 100 (death)) at 90 days after the surgical intervention
Correlation between preoperative anxiety and preoperative Patient Health Engagement Scale (PHE-S) | From 14 days to 1 day before surgery
  Correlation between preoperative anxiety- assessed through the Hospital Anxiety and Depression Scale (HADS) (Self-reported scale ranging from 0 to 21, where significant anxiety and depression are identified by a 8 point cut-off) and the preoperative Patient Health Engagement Scale (PHE-S, self-reporting scale ranging from 0 (complete disease awareness) to 12 (complete absence of disease awareness).
Correlation between preoperative anxiety and C-Reactive Protein (CRP) level 24 hour after surgery | 24 hours after surgery
  Correlation between preoperative anxiety- assessed through the Hospital Anxiety and Depression Scale (HADS) (Self-reported scale ranging from 0 to 21, where significant anxiety and depression are identified by a 8 point cut-off) and the level of serum C-Reactive Protein (CRP, µg/mL) measured 24 hours after surgery.
90-day postoperative complications | 90 days after surgery
  Rate difference of 90-day postoperative complications (classified according to the Clavien-Dindo scale) between the interventional cohort and the historical cohort of comparison.
Correlation between the 90-day Postoperative Recovery Profile (PRP) and 90-day Heart Rate Variability (HRV) | 90 days after surgery
  Correlation between the 90-day Postoperative Recovery Profile (PRP) (Scale ranging from 0 (completely recovered) to 68 (not recovered)) and the median value of at least twelve Heart Rate Variability (HRV) measures collected in the postoperative period through the Howdy Senior® device.
Healthcare costs | 6 months after surgery
  Median difference of the healthcare resources used in the interventional cohort and the historical cohort of comparison.

CONTACTS AND LOCATIONS:
Overall Officials: Antonino Spinelli, MD, PhD, Principal Investigator — IRCCS Huamanitas Research Hospital
Locations (1):
- IRCCS Humanitas Research Hospital, Rozzano, MI, Italy

IPD SHARING:
Plan to Share IPD: No